CLINICAL TRIAL: NCT05340790
Title: A Phase 1 Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of Antimicrobial Peptide PL-18 Vaginal Suppositories in Healthy Adult Subjects
Brief Title: First in Human Study in Healthy Volunteers of Antimicrobial Peptide PL-18 Vaginal Suppositories
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Protelight Pharmaceuticals Australia PTY LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JSPL-PL-18-101
Record Dates: First submitted 2022-02-23; First posted 2022-04-22 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Colpomycosis; Bacterial Vaginosis; Mixede Vaginitis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antimicrobial Peptide PL-18 Vaginal Suppositories (Experimental): Dose 1 to 5 of Antimicrobial Peptide PL-18 Vaginal Suppositories
  Interventions: Drug: Dose 1 to 5 of Antimicrobial Peptide PL-18 Vaginal Suppositories
- Placebo dose (Placebo Comparator): Placebo dose 1 to 5 of Antimicrobial Peptide PL-18 Vaginal Suppositories
  Interventions: Drug: Placebo dose 1 to 5 of Antimicrobial Peptide PL-18 Vaginal Suppositories

INTERVENTIONS:
Drug: Dose 1 to 5 of Antimicrobial Peptide PL-18 Vaginal Suppositories — Escalating doses of 1 mg (0.1%)、2.5mg (0.25%)、5 mg (0.5%)、10mg (1%)、15 mg (1.5%)；single dose administration；topical vaginal suppository ；multiple-dose administration after single dose administration a 3-day wash out period ; once-daily for 6 consecutive days;
  Other Names: AMP PL-18
  Arms: Antimicrobial Peptide PL-18 Vaginal Suppositories
Drug: Placebo dose 1 to 5 of Antimicrobial Peptide PL-18 Vaginal Suppositories — Dose 1、2、3、4 and 5 of Antimicrobial Peptide PL-18 Vaginal Suppositories respective placebos；single dose administration；topical vaginal suppository ；multiple-dose administration after single dose administration a 3-day wash out period ; once-daily for 6 consecutive days;
  Other Names: Placebo PL-18
  Arms: Placebo dose

SUMMARY:
This is a Single-center, Randomized, Double-blind, Placebo-controlled Phase I Study to Evaluate the Safety, Tolerability and PK Profiles of Single and Multiple Ascending Doses of Antimicrobial Peptide PL-18 Vaginal Suppositories.

DETAILED DESCRIPTION:
Subjects who provide written informed consent to participate voluntarily in the clinical study will be screened. Eligible subjects will be sequentially enrolled into the above five sequential cohorts and randomized to receive PL-18 (cohort 1: n=8; cohort 2/3/4/5: n=6) or matching placebo (n=2). Subjects will be observed for 3 days after a single dose and receive PL-18 or placebo, once daily, for 6 consecutive days, if no grade ≥2 drug-related adverse events (AEs) occur. During the study, PK sample collection, physical examination, vital signs, laboratory tests, electrocardiography (ECG) and tolerance evaluation will be performed based on the protocol schedule.

To ensure the safety of the subjects, two sentinel subjects will be enrolled first in each cohort; one subject will be randomized to receive PL-18, and the other subject randomized to receive placebo. The safety data of the two sentinel subjects from initiation of single dosing to the last drug administration of multiple dosing on D11 will be reviewed by the investigator and sponsor before the subsequent subjects in that dose cohort are enrolled. Subsequent subjects could be simultaneously enrolled, with one randomized to receive placebo and others randomized to receive PL-18.

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for inclusion in this study only if all of the following criteria are met:

  1. Voluntarily signed written informed consent;
  2. Ability to comprehend the purpose of the study; ability to co-operate with the investigator and comply with all study requirements;
  3. Adult females aged between 18 and 55 years (inclusive);
  4. Body weight between 50 and 100 kg (inclusive) and body mass index (BMI) within 18~32 kg/m2 (inclusive).
  5. In good health as determined by screening tests. Good health is defined as having no clinically relevant abnormalities identified by a detailed medical history, full physical examination (including measurement of blood pressure and pulse rate), 12-lead ECG, and clinical laboratory tests:

     * Vital signs (measured after resting for 5 minutes seated position) within normal range, or outside the normal range and not considered clinically significant by the Investigator;
     * Standard 12-lead ECG parameters (recorded after resting for 5 minutes in supine position) in the following ranges; QTc (Fridericia algorithm recommended) ≤470 ms, and normal ECG tracing, or abnormal ECG tracing not considered clinically relevant by the Investigator;
     * Laboratory parameters demonstrating no clinically significant abnormalities, as determined by the Investigator. A total bilirubin outside the normal range may be acceptable if total bilirubin does not exceed 1.5 × ULN conjugated bilirubin (with the exception of a participant with documented Gilbert syndrome).
  6. Self-report regular menstrual cycle (21-35 days), and planned to avoid menstruation from the first administration until 7 days after the last administration;
  7. Negative human papilloma virus (HPV) test result (at screening or negative HPV test result performed in study site within 2 months prior to screening;
  8. History of sexual life, including vaginal intercourse;
  9. Be willing to use vaginal suppositories;
  10. Currently in a mutually monogamous sexual relationship or no sexual activity;
  11. Sexual abstinence from 72 hours prior to the first drug administration until 7 days after the last administration;
  12. Agreement to avoid the use of any other intravaginal products (i.e., contraceptive creams, gels, foams, sponges, lubricants, irrigation solutions, etc.) from screening until 7 days after the last administration;
  13. Subjects in a intercourse relationship must agree to use highly effective methods of contraception (as specified in Section 4.6.3) from informed consent obtained until 3 months after the last administration, and pregnancy test results must be negative at screening.

Exclusion Criteria:

* A subject meeting any of the following exclusion criteria will not be allowed to participate in this study:

  1. Significant deep epithelial disruption by colposcopy at screening;
  2. Anatomical anomalies of the genito-urinary tract and vaginal prolapse;
  3. Genitourinary infections at screening or within 21 days prior to screening, including but not limited to bacterial urinary tract infection, bacterial vaginosis, trichomoniasis and vulvovaginal candidiasis;
  4. Known, active sexually transmitted infection (STI) in partner, as per anamnesis;
  5. Two or more confirmed trichomoniasis, gonococcal, chlamydia trachomatis or syphilis spirochete infections within 180 days prior to screening;
  6. History of recurrent genital herpes or active herpes simplex virus (HSV) at screening;
  7. Hepatitis B virus, hepatitis C virus, human immunodeficiency virus (HIV), syphilis infection, or positive hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C virus antibody (HCVAb), HIV antibody (HIVAb), treponema pallidum antibody (TP-Ab) at screening;
  8. History of clinically severe relevant cardiovascular, hepatic, renal, pulmonary, gastrointestinal, endocrine, or neurological diseases that, in the investigator's opinion, may interfere with the aim of the study or affect the subject's safety;
  9. Uncontrolled or acute illness that may complicate the study evaluation in the investigator's opinion;
  10. History of hysterectomy;
  11. Pelvic surgery within 90 days prior to screening;
  12. Cervical cryotherapy or cervical laser treatment within 90 days prior to screening;
  13. Intrauterine device insertion or removal within 90 days prior to screening;
  14. Any antibiotic or antifungal therapy (intravaginal or systemic) within 30 days prior to screening;
  15. Immunosuppressive therapy within 60 days prior to screening;
  16. Ascertained or presumptive hypersensitivity (including allergies) to any ingredient of the investigational medicinal product (IMP); history of other significant anaphylaxis to drugs or allergic reactions in general;
  17. Pregnant or lactating women, or women within 60 days of the last pregnancy;
  18. Subjects who consume or are unable to abstain from products containing caffeine/xanthine within 24 hours before a visit or admission;
  19. History of drug or alcohol abuse within 1year prior to screening, or a positive result of drug abuse or alcohol breath test at screening or check-in;
  20. Previously dosed with an investigational drug within 3 months prior to Day 1 or still participating in another trial at the time of screening;
  21. Any vaccination from the 28 days prior to administration of the first dose until 28 days after the last dose;
  22. Those considered by the investigator as inappropriate to participate in the study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Characterize safety profile of Antimicrobial Peptide PL-18 Vaginal Suppositories about the incidence of treatment emergent adverse events | 38 days
  All AEs will be summarized by system organ class (SOC) and preferred term (PT). The numbers and percentages of subjects experiencing AEs will be calculated.
The numbers and percentages of subjects experiencing vital sign abnormalities with/without clinical significance. | 17 days
  Vital signs abnormalities will be summarized with descriptive statistics. Vital signs include body temperature, blood pressure, heart rate/pulse, respiration. Changes from the baseline of each test over time will be summarized.
The numbers and percentages of subjects experiencing physical examination abnormalities with/without clinical significance. | Day 4 , Day 11 , Day 17
  Physical examinations abnormalities will be summarized with descriptive statistics. Physical examination will include general condition, skin, head, eyes, ears, nose, throat, heart, lungs, chests, abdomen, extremities, nerves, back/spine, lymph, nodes. Changes from the baseline of each test over time will be summarized.
Safety assessment about the changes of clinical laboratory tests. | Day2, Day 4 , Day5, Day 8, Day 11 , Day 17
  Laboratory abnormalities will be summarized with descriptive statistics. Clinical laboratory tests include hematology, blood chemistry, level of immune factors, urinalysis.
Safety assessment about the changes of 12-lead ECG . | Day1, Day 4 , Day 5, Day 7, Day 11 , Day 17
  12-lead ECG abnormalities will be summarized with descriptive statistics.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Day1~Day4
  Concentrations of Antimicrobial Peptide PL-18 in Plasma samples at different time points are measured.Maximum plasma concentration (Cmax) is a PK parameter of the single-dose stage.Plasma concentrations at different time points will be listed and summarized by descriptive statistics.
Time to Maximum plasma concentration (Tmax) | Day1~Day4
  Tmax is a PK parameter of the single-dose stage.Plasma PK parameters will be analyzed by non-compartmental analysis (NCA) with WinNonlin® version 8.1 or above and SAS® version 9.4 or higher.
Area under the concentration-time curve from the time zero to last measurable concentration (AUC0-t) | Day1~Day4
  AUC0-t is a PK parameter of the single-dose stage.Plasma PK parameters will be analyzed by non-compartmental analysis (NCA) with WinNonlin® version 8.1 or above and SAS® version 9.4 or higher.
Area under concentration-time from time zero to infinity (AUC0-inf) | Day1~Day4
  AUC0-t is a PK parameter of the single-dose stage.Plasma PK parameters will be analyzed by non-compartmental analysis (NCA) with WinNonlin® version 8.1 or above and SAS® version 9.4 or higher.
Terminal half-life (t1/2) | Day1~Day4
  t1/2 is a PK parameter of the single-dose stage.Plasma PK parameters will be analyzed by non-compartmental analysis (NCA) with WinNonlin® version 8.1 or above and SAS® version 9.4 or higher.
Apparent clearance (CL/F) | Day1~Day4
  CL/F is a PK parameter of the single-dose stage.Plasma PK parameters will be analyzed by non-compartmental analysis (NCA) with WinNonlin® version 8.1 or above and SAS® version 9.4 or higher.
Apparent volume of distribution (Vz/F) | Day1~Day4
  Vz/F is a PK parameter of the single-dose stage.Plasma PK parameters will be analyzed by non-compartmental analysis (NCA) with WinNonlin® version 8.1 or above and SAS® version 9.4 or higher.
Mean residence time (MRT) | Day1~Day4
  MRT is a PK parameter of the single-dose stage.Plasma PK parameters will be analyzed by non-compartmental analysis (NCA) with WinNonlin® version 8.1 or above and SAS® version 9.4 or higher.
Terminal elimination rate constant (λz) | Day1~Day4
  λz is a PK parameter of the single-dose stage.Plasma PK parameters will be analyzed by non-compartmental analysis (NCA) with WinNonlin® version 8.1 or above and SAS® version 9.4 or higher.
Maximum observed concentration at steady state (Cmax,ss) | Day5~Day 11
  Concentrations of Antimicrobial Peptide PL-18 in Plasma samples at different time points are measured.Maximum observed concentration at steady state (Cmax,ss) is a PK parameter of the multi-dose stage.
Minimum observed concentration at steady state (Cmin,ss) | Day5~Day 11
  Concentrations of Antimicrobial Peptide PL-18 in Plasma samples at different time points are measured. Minimum observed concentration at steady state (Cmin,ss) is a PK parameter of the multi-dose stage.
The average concentration during a dosing interval at steady state (Cav,ss) | Day5~Day 11
  The average concentration during a dosing interval at steady state (Cav,ss) is a PK parameter of the multi-dose stage. Plasma PK parameters will be analyzed by non-compartmental analysis (NCA) with WinNonlin® version 8.1 or above and SAS® version 9.4 or higher.
Area under the concentration-time curve from zero to the end of the dosing interval at steady state (AUCss) | Day5~Day 11
  AUCss is a PK parameter of the multi-dose stage. Plasma PK parameters will be analyzed by non-compartmental analysis (NCA) with WinNonlin® version 8.1 or above and SAS® version 9.4 or higher.
Accumulation ratio (Rac) | Day5~Day 11
  Accumulation ratio (Rac) is a PK parameter of the multi-dose stage. Plasma PK parameters will be analyzed by non-compartmental analysis (NCA) with WinNonlin® version 8.1 or above and SAS® version 9.4 or higher.
Characterize the effect of Antimicrobial peptide PL-18 Vaginal Suppositories on vaginal bacteria | 17 days
  Changes in vaginal bacteria after single and multiple doses of Antimicrobial Peptide PL-18 Vaginal Suppositories in healthy adult female subjects assessed. Changes in vaginal bacteria will be summarized with descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: John McNeil, Professor, Study Chair — 90768825
Locations (1):
- Q-Pharm Pty. Ltd, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No